CLINICAL TRIAL: NCT02353702
Title: Efficacy of Parietal Continuous Infiltration of Local Anesthesic on Diaphragmatic Function After Upper Abdominal Surgery Through a Subcostal Incision
Brief Title: Efficacy of Local Anesthesic on Diaphragmatic Function After Upper Abdominal Surgery
Acronym: CATPAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012/176/HP
Record Dates: First submitted 2015-01-22; First posted 2015-02-03 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Hepatectomy
Keywords: Diaphragmatic function; sniff-test; pulmonary complications; upper abdominal surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infusion of Ropivacaine during 48 hours (Experimental): Evaluation of diaphragmatic function with Sniff test after 48h continuous parietal infiltration of Ropivacaine using parietal catheter at the following dose :
  20 ml Bolus (7,5 mg/ml) then continuous administration of 10 ml per hour (2 mg/ml)
  Interventions: Procedure: Sniff test; Drug: Infusion of Ropivacaine during 48 hours; Device: Continuous parietal infusion with parietal catheter; Drug: NaCl
- Infusion of placebo during 48 hours (Placebo Comparator): Evaluation of diaphragmatic function with Sniff test after 48h continuous parietal infiltration of placebo using parietal catheter at the following dose :
  20 ml Bolus (NaCl 0.9 %) then continuous administration of 10 ml per hour (NaCl 0.9 %)
  Interventions: Procedure: Sniff test; Device: Continuous parietal infusion with parietal catheter; Drug: Infusion of placebo during 48 hours; Drug: NaCl

INTERVENTIONS:
Procedure: Sniff test — Evaluation of diaphragmatic function by sniff test after continuous parietal infusion of ropivacaine or placebo
Drug: Infusion of Ropivacaine during 48 hours — 20 ml Bolus (7,5 mg/ml) then continuous administration of 10 ml per hour (2 mg/ml) during 48 hours of Ropivacaine.
  20 ml Bolus (NaCl 0.9 %) then continuous administration of 10 ml per hour, during 48 hours of NaCl 0.9 %.
  Arms: Infusion of Ropivacaine during 48 hours
Device: Continuous parietal infusion with parietal catheter — Continuous parietal infiltration of Ropivacaine or placebo
Drug: Infusion of placebo during 48 hours
  Arms: Infusion of placebo during 48 hours
Drug: NaCl

SUMMARY:
Upper abdominal surgery is known to induce such pulmonary complications as pneumonia, atelectasis, pleural effusion. The post operative diaphragmatic dysfunction participates to these complications and lasts for 7 days after upper abdominal surgery. The sniff-test is a recognized tool for measuring the diaphragmatic function.The purpose of this study is to evaluate the effectiveness of parietal analgesia with continuous infiltration of local anesthesic on diaphragmatic function after upper abdominal surgery through a subcostal incision. Our main outcome is to measure the diaphragmatic function with the sniff test in 44 patients with parietal infiltration of ropivacaine and in 44 patients with placebo. Our secondary outcomes are the evaluation of the effect of continuous parietal analgesia with ropivacaine on IPmax and EPmax, oxygen saturation, post operative pulmonary complications and post operative recovery. This prospective study will determine if the pre peritoneal local infiltration of ropivacaine is useful to decrease post operative diaphragmatic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Surgical Indication for Upper abdominal surgery through subcostal incision
* More than 18 years old , less than 80 years old
* ASA score between 1 and 3
* Effective contraception for more than 3 months in women of childbearing age
* Patients signed an informed consent
* Affiliation to a social security regimen

Exclusion Criteria:

* BMI more than 30 kg/m2
* Nasal obstruction during inclusion
* Preoperative treatment with morphine
* Need for a postoperative nasogastric tube
* Difficulty to understand the use of the PCA and/or the sniff-test
* Impossibility to place the catheter in preperitoneal position
* Pregnant women or breasting women
* Patients under guardianship
* Contraindication to use of ropivacaine
* Inclusion in another clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Buccal Inspiratory Pression (IP) Evaluation of diaphragmatic function using sniff test. | Day 6 post surgery
  Evaluation of diaphragmatic function using sniff test. The measured value is buccal inspiratory pression.

SECONDARY OUTCOMES:
Maximal buccal inspiratory pression (IPmax) using sniff test | Day 6 after surgical procedure
  Evaluation of maximal buccal inspiratory pression (IPmax) using sniff test
Maximal buccal expiratory pression (EPmax) using sniff test | Day 6 after surgical procedure
  Evaluation of maximal buccal expiratory pression (EPmax) using sniff test
Oxygen saturation rate | Day 6 after surgical procedure
  Evaluation of Oxygen saturation
medical complication outcome (pneumonia) | week 6 after surgical procedure
  Medical pulmonary complications outcome : pneumonia
medical complication outcome (atelectasis) | week 6 after surgical procedure
  Medical pulmonary complications outcome : atelectasis
medical complication outcome (pleural effusions) | week 6 after surgical procedure
  Medical pulmonary complications outcome : pleural effusions
Morphine consummation (Measurement of Morphine consummation since surgery) | week 6 after surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Michel SCOTTE, Pr, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France